CLINICAL TRIAL: NCT04994171
Title: Operative Difficulty Grading Scale for Laparoscopic Cholecystectomy in BPKIHS
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Nirmal Prasad Sah, Assistant Professor, B.P. Koirala Institute of Health Sciences
Other Study IDs: 1758/020
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Surgery; Laparoscopic; Cholecystectomy; Cholecystitis
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of this study is to utilize operative grading scale to predict conversion to open,complication and reintervention and validate Nassar Scale.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is the commonly performed procedure in our institute. Laparosopic cholecystectomy is high variable surgery ranging from simple routine operation to difficult surgery leading to increased morbidity and mortality. The majority of previous scores use a combination of pre-operative and operative data and were produced in studies that were limited by retrospective data, small sample sizes and lack of external validation.

Very few intraoperative difficulty grading scale was published and none are widely used in clinical practice. So operative grading scale will have advantages of assisting in intra-operative strategy and planning, allowing comparison across different research studies, facilitating risk adjustment for surgical outcomes and providing an aid in training surgeons and monitoring of training progression.

The main purpose of this study is to utilize operative grading scale to predict conversion to open,complication and reintervention.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing laparoscopic cholecystectomy

Exclusion Criteria:

* CBD Stone
* Malignancy of Extrahepatic biliary tree
* Cholecystectomy as a part of other surgery

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hospital patients
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Laproscopic cholecystectomy Conversion to open with Nassar Grade | 30 day
  Laproscopic cholecystectomy converted to open with Nassar grade ie chance of conversion to open in higher Nassar grade(difficult laparoscopic cholecystectomy)
Duration of Surgery | 30 day
Introperative Complication with Nassar Grade | 30 day
  Complication like biliary spillage, stone spillage and bleeding with higher Nassar grade (difficult laparoscopic cholecystectomy)

SECONDARY OUTCOMES:
Total length of stay | 30 day

CONTACTS AND LOCATIONS:
Locations (1):
- Nirmal Prasad sah, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandio A, Timmons S, Majeed A, Twomey A, Aftab F. Factors influencing the successful completion of laparoscopic cholecystectomy. JSLS. 2009 Oct-Dec;13(4):581-6. doi: 10.4293/108680809X1258998404560. PMID 20202401
- [Background] Ahmed N, Hassan MU, Tahira M, Samad A, Rana HN. Intra-Operative Predictors of difficult cholecystectomy and Conversion to Open Cholecystectomy - A New Scoring System. Pak J Med Sci. 2018 Jan-Feb;34(1):62-66. doi: 10.12669/pjms.341.13302. PMID 29643880
- [Result] Jameel SM, Bahaddin MM, Mohammed AA. Grading operative findings at laparoscopic cholecystectomy following the new scoring system in Duhok governorate: Cross sectional study. Ann Med Surg (Lond). 2020 Oct 23;60:266-270. doi: 10.1016/j.amsu.2020.10.035. eCollection 2020 Dec. PMID 33204417